CLINICAL TRIAL: NCT04789863
Title: Towards Implementation of an Integrated Model of Care in Long-Term Follow-Up After Allogeneic Hematopoietic SteM Cell TransplantatIon faciLitated by eHealth Technology (The SMILe Project) - An Effectiveness-implementation Science Study
Brief Title: Implementation and Testing of an eHealth Integrated Model of Care for Patients Receiving Allogeneic Stem Cell Transplantation: The SMILe Project
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Basel (Other)
Collaborators: University Hospital Freiburg (Other); University Hospital, Basel, Switzerland (Other); University of Applied Science Augsburg, Germany (Unknown); KU Leuven (Other); University Hospital, Zürich (Other); University Hospital, Geneva (Other)
Responsible Party: Principal Investigator, Sabina De Geest, Prof. Dr.; PhD, RN, FAAN, FRCN, FEANS, University of Basel
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: SMILe
Record Dates: First submitted 2021-03-03; First posted 2021-03-10 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: Stem Cell Transplantation
Keywords: Implementation Science; Delivery of Health Care, Integrated; Telemedicine; Advanced Practice Nursing; Randomized Controlled Trial; Self-Management

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention group (Other): Intervention group (IG) patients will receive usual care plus the SMILe-ICM (see below) when they come to their planned follow-up appointments at the University Hospital Basel. Thus, while IG participants will receive the same number of follow-up appointments as CG participants (depending on their state of health), they will also receive the SMILe-ICM, i.e., tailored self-management and behavioural support delivered by the combination of totally 12 face-to-face meetings with a Care Coordinator (CC) and the SMILeApp. The personal meetings with the CC will last around 40-90 minutes. The first three of them will occur during the initial alloSCT hospitalization, and the other nine will occur in the outpatient setting, beginning with biweekly and expanding to bi-monthly intervals until one year post-alloSCT.
  Interventions: Device: SMILe-Integrated Care Model
- Control group (Other): see "Intervention" section
  Interventions: Other: Usual Care

INTERVENTIONS:
Device: SMILe-Integrated Care Model — Four self-management intervention modules will be delivered by human and technology: 1) monitoring & follow-up; 2) infection prevention; 3) medication adherence; 4) physical activity.
  Human. A CC will provide structured and tailored self-management and behavioural support regarding all 4 modules via 12 face-to-face meetings congruent with planned clinic follow-up visits. The CC will be connected with the patients via the SMILe technology, enabling rapid responses to early signs of health deterioration.
  Technology. The SMILe technology consists of the SMILeApp and SMILeCare. The latter is the interface of the monitoring component to connect the patient with the CC supporting fast recognition of symptoms and health deterioration. The SMILeApp enables to daily record a set of medical, behavioural and symptom-related data. A lexicon provides self-management and behavioural information. All data will be transferred to the clinic to be monitored, with the patient's consent, via SMILeCare.
  Arms: Intervention group
Other: Usual Care — The control group (CG) participants will receive usual care, which includes no specific counselling. USB outpatient appointment frequency follows a standard schedule: during the first 3 months post-alloSCT, depending on their health status, most patients (73%) return 1 to 3 times per week for follow-up at the USB outpatient clinic, where they are mainly seen by a junior or senior physician. Depending on health status and recovery, follow-up intervals extend to weekly or monthly within 1 year post-alloSCT. A research assistant (RA) will just contact CG participants for data collection. If participants raise concerns about any symptoms, the RA will encourage them to contact their physicians.
  Arms: Control group

SUMMARY:
Numerous publications call for innovation based on integrated care principles, investment in self-management and use of eHealth to improve outcomes for allogeneic Stem Cell Transplant (alloSCT). While eHealth supported integrated care models are effective, real-world implementation remain elusive.

The newly developed SMILe-Integrated Care Model (ICM) is the first theory-based eHealth supported integrated care model for alloSCT patients. SMILe-ICM includes four self-management modules (i.e., monitoring & follow-up, medication adherence, infection prevention, physical activity) and combines a human role, i.e., a Care Coordinator (CC), with a technological component (i.e., the SMILeApp). Patients monitor and transfer symptoms and health behaviours to their CC, who supports them in self-management and dealing with complications.

Embedded in implementation science methodology, we aim to implement and test the SMILe-ICM at the University Hospital Basel (USB) in the first year post-alloSCT by evaluating effectiveness, implementation outcomes and implementation pathway.

A hybrid 1 effectiveness-implementation randomized controlled trial will include 80 adult alloSCT patients who are transplanted and followed up at USB, have basic German proficiency and provide written informed consent. Patients with physical or mental conditions limiting the use of the SMILeApp will be excluded. About ten days before alloSCT, a stratified randomization based on participants' clinical risk scores will assign patients 1:1 to the control (CG) or intervention group (IG). The CG will receive usual care; the IG will receive the SMILe-ICM over one year with 12 CC visits and continuous use of the SMILeApp. Re-hospitalization rate (primary outcome), total healthcare utilization costs, acute and chronic GvHD episodes and survival will be assessed using medical records. Medication adherence will be assessed via the BAASIS© scale, treatment burden via the PETS©, health-related quality of life via the EQ-5D-5L©. Implementation outcomes will be assessed via questionnaires and the implementation pathway via qualitative focus groups, each from patient and CC perspectives. Patients will be followed up 3 months after the intervention ended. Intention-to-treat and per-protocol analyses will be conducted using the rate ratio by unconditional maximum likelihood estimation (Wald) for the primary outcome. Qualitative data will be analysed using mind-mapping techniques and thematic analysis.

DETAILED DESCRIPTION:
Background. Numerous publications call for innovation based on integrated care principles, investment in self-management and use of eHealth to improve outcomes for allogeneic Stem Cell Transplant (alloSCT), patients with complex care needs and multiple morbidities. While eHealth supported integrated care models are effective, real-world implementation and sustainability remain elusive. Combining implementation science with computer and behavioural science methods, we will implement and evaluate the newly developed SMILe-Integrated Care Model (SMILe-ICM) for alloSCT patients, aiming to reduce first year post-alloSCT re-hospitalizations.

The SMILe-ICM is the first theory-based comprehensive eHealth supported integrated care model. Developed by marrying different methodological approaches, it comprehensively addresses alloSCT needs by optimizing care coordination and care processes, and by reducing response times in cases where the patient's condition is deteriorating at home. SMILe-ICM includes four self-management care modules (i.e., monitoring & follow-up, medication adherence, infection prevention, physical activity) and combines a human role newly embedded in the SCT team, i.e., a Care Coordinator (CC), with a technological component (i.e., the SMILeApp). Patients' symptoms and health behaviours are monitored and transferred, as necessary, to their CC, who supports them in their self-management. Alongside the alloSCT team, the CC manages complications based on care algorithms. Thus, SMILe-ICM targets alloSCT patients' clinical and behavioural short- (e.g., infections) and medium-term outcomes (e.g., adherence, treatment burden, GVHD). Our SMILe-ICM pilot work indicates high-level acceptability, feasibility and technological performance.

Purpose. Embedded in implementation science methodology, we aim to implement and test the SMILe-ICM at the University Hospital Basel (USB) in the first year post-alloSCT. In addition to targeting one primary outcome, re-hospitalization rate, our secondary outcomes will include effectiveness (e.g., health care costs, medication adherence) and implementation outcomes (e.g., acceptability, fidelity). We will also describe and evaluate our implementation pathway. Patients will be followed up 3 months after the end of the intervention period.

Methods. A hybrid 1 effectiveness-implementation randomized controlled trial will include 80 adult alloSCT patients from the USB Department of Haematology who are transplanted and followed up at USB, have basic German proficiency and elementary computer literacy, and who provide written informed consent. Patients with physical or mental conditions limiting their use of the SMILe-ICM's technology component will be excluded. Approximately ten days before the scheduled alloSCT, a stratified randomization (based on participants' clinical risk scores) will assign patients 1:1 to the control group (CG) or the SMILe-ICM intervention group (IG). The CG will receive usual care; the IG will receive the SMILe-ICM (see above) over one year with 12 scheduled CC visits and continuous use of the SMILeApp. The re-hospitalization rate (primary outcome) and total healthcare utilization costs (payers' perspective) will be assessed using medical records. Medication adherence will be assessed via the BAASIS© scale, treatment burden via the PETS© scale, health-related quality of life via the EQ-5D-5L© (value set for Germany EQ-VT v. 2.0-quality-adjusted life years), and acute and chronic GvHD episodes and survival via medical records. Implementation outcomes will be assessed from both patient and CC perspectives via questionnaires and the implementation pathway via qualitative data collection techniques (i.e., focus groups with patients, clinicians). Quantitative data will be collected using a blinded standardized method in patients' first year post-alloSCT, then 3 months thereafter. Intention-to-treat and per-protocol analyses will be conducted using the rate ratio by unconditional maximum likelihood estimation (Wald) for the primary outcome. Qualitative data will be analysed using mind-mapping techniques and thematic analysis.

Conclusion: The SMILe-ICM implies a systemic innovation in the follow-up care of alloSCT patients, targeting short- and medium-term outcomes. Bolstering patient's self-management, this eHealth-supported behavioural science-driven integrated care approach aims at fast responses to health deterioration. This implementation science methodological innovation will also develop insights regarding the implementation process. Should it prove effective, then, it will also prepare the SMILe-ICM for scaling up or out to other chronically ill patient populations.

ELIGIBILITY:
Inclusion Criteria:

* Patient's allogeneic stem cell transplantation and follow-up treatment is planned at the University Hospital Basel
* Aged ≥ 18 years
* Able to speak, read and write German at least limited working proficiency (i.e., to satisfy conversations and understand written material regarding routine social demands and limited requirements)
* Able to plan and perform self- management activities independently
* WLAN access at home or own a sufficient mobile data contract
* Normal, mental, physical and psychological abilities and health to provide a written informed consent about study participation and related data protection

Exclusion Criteria:

* General condition make self-management impossible for more than 4 weeks
* Follow up care solely at an external center
* Diagnosed with dementia
* A second allogeneic stem cell transplantation becomes necessary

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2023-10-31 (Actual); Study Completion 2023-10-31 (Actual)

PRIMARY OUTCOMES:
Change of re-hospitalization rate from post-alloSCT discharge up to 15 months after allogeneic stem cell transplantation | Data will be collected monthly via medical records during the study period, i.e., until one year post-alloSCT and for a further period of 3 months to test for a possible wane out effect.
  The number of events after the initial post-alloSCT discharge per patient

SECONDARY OUTCOMES:
Change of total healthcare utilization costs from post-alloSCT discharge until 15 months post-alloSCT | Data will be collected monthly during the study period, i.e., until one year post-alloSCT and for a further period of 3 months to test for a possible wane out effect.
  Will be calculated from the payers' perspective, i.e., based on type of insurance (public/private), standardized unit costs of resources in Switzerland, and medical records. Costs for 5 healthcare utilization classes will be counted: physician visits, ambulatory healthcare visits, rehabilitation services, home care services, inpatient days. Information about home care services is not available via medical records and will be obtained via an adapted version of the FIMA© self-reporting questionnaire. For this study, the FIMA© was shortened to 7 items, asking retrospectively for number of physicians visits, d/hrs of ambulatory healthcare visits, d/hrs of home care services, d/hrs of support by family caregivers, type & duration of rehabilitation therapy, reason & duration of inpatient days, type of insurance. Comparing the data collected via the FIMA© will check the data validity of medical records. In case of incongruences, valid data from medical records will be used.
Change of medication adherence from post-alloSCT discharge until 15 months post-alloSCT | Data will be collected monthly (BAASIS©) and daily (MEMS® Button) during the study period as long as patients need to take immunosuppressants, i.e., at the longest until 1 year post-alloSCT and for a further period of 3 months.
  Medication non-adherence (implementation & persistence dimension) will be assessed using the Basel Assessment of Adherence to Immunosuppressive Medication Scale (BAASIS©).The BAASIS© is a validated self-report measure assessing adherence to implementation issues (e.g., drug holidays; 4 items; YES/NO) and persistence/discontinuation (1 item; Yes/No). In addition, we will apply electronic monitoring (EM), i.e., the MEMS® Button, an electronic pillbox system recording the date and time of each medication intake. As described in our previous MAESTRO-TX study, the electronically compiled dosing history will be expressed as a sequence of daily binary adherence scores per patient.
Change of treatment burden from baseline until 12 months post-alloSCT | Data will be collected at baseline, days +90, +180 and +365 via self-report questionnaire (PETS©) during the intervention period.
  Treatment burden will be measured via the German version of the PETS© self-reporting questionnaire. This includes nine multi-item domain scales, each measuring the burden of one aspect of chronic illness treatment: medical information (7 items); medications (7 items); medical appointments (3 items); health monitoring (2 items); interpersonal challenges (4 items); health care expenses (5 items); difficulty with health care services (7 items); role/social activity limitations due to self-management (6 items); and physical/mental exhaustion due to self-management (5 items). Items apply 4- or 5-point Likert-type response scales regarding a 4-week recall time frame. Raw domain scores are transformed to a standardized 0-to-100 metric, with higher scores indicating greater treatment burden.
Change of HRQL from baseline until 12 months post-alloSCT | Data will be collected monthly via medical records during the intervention period, i.e., until one year post-alloSCT.
  HRQL will be measured using the EQ-5D-5L©,a validated instrument covering five dimensions (mobility, self-care, usual activities, pain/discomfort and anxiety/depression) and including the EQ-Visual Analogue Scale (VAS), on which individuals rate their overall perceived health state (scale of 0 to 100).
Change of QALY from baseline until 12 months post-alloSCT | Data will be collected monthly during the intervention period, i.e., until one year post-alloSCT.
  We will also calculate quality-adjusted life years (QALY), as QALY scores are required for the National Institute for Health and Clinical Excellence (NICE) health technology assessment. As a standardized measure of disease burden which combines both survival and health-related quality of life into a single index, the QALY scores provide a 'common currency' of comparison across disease areas. Generating them requires the preference weight of HRQL (obtained from the EQ-5D-5L© value set for Germany EQ-VT v. 2.0) and time between each HRQL measurement. QALY scores range from 1 (perfect health) to 0 (dead).
Change of GvHD from post-alloSCT until 12 months post-alloSCT | Data will be collected monthly during the intervention period, i.e., until one year post-alloSCT.
  Incidence and grade of chronic and acute GvHD will be retrieved from medical records.
Change of implementation outcomes and process evaluation from baseline until 15 months post-alloSCT | Data will be collected monthly via medical records during the study period, i.e., until one year post-alloSCT and for a further period of 3 months to test for a possible wane out effect.
  Overall survival rate will be retrieved from medical records.
Change of overall survival rate from post-alloSCT until 15 months post-alloSCT | Data will be collected via medical records at days +30, +60, +90, +120, +150, +180, +240, +300, +365 and +455
  Overall survival rate after having received the alloSCT
Patient's demographics at baseline | At baseline: 10 days before alloSCT
  Patient's demographics will be assessed as follows: age, sex, education, living alone
Patient's clinical characteristics at baseline | At baseline: 10 days before alloSCT
  Patient's clinical characteristics will be assessed as follows: conditioning regimen, donor match/type, disease status at transplant, time diagnosis to transplant

CONTACTS AND LOCATIONS:
Overall Officials: Sabine De Geest, Prof., Principal Investigator — Nursing Science, Department Public Health, University of Basel, Switzerland
Locations (1):
- University Hospital Basel, Basel, Basel, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] De Geest S, Valenta S, Ribaut J, Gerull S, Mielke J, Simon M, Bartakova J, Kaier K, Eckstein J, Leppla L, Teynor A; SMILe team. The SMILe integrated care model in allogeneic SteM cell TransplantatIon faciLitated by eHealth: a protocol for a hybrid effectiveness-implementation randomised controlled trial. BMC Health Serv Res. 2022 Aug 20;22(1):1067. doi: 10.1186/s12913-022-08293-8. PMID 35987671